CLINICAL TRIAL: NCT01275846
Title: Study for Deployment of American Heart Association Heart Failure Protocols and Educational Content Within the Intel® Health Guide System With a Congestive Heart Failure Cohort
Brief Title: Deployment of American Heart Association Heart Failure Protocols and Content Within the Intel® Health Guide System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Heart Association (Other)
Collaborators: Intel Corporation (Industry)
Responsible Party: Principal Investigator, Ileana L. Piña, Professor of Medicine & Epidemiology and Population Health, Albert Einstein College of Medicine, Montefiore Medical Center, American Heart Association
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AHA100602; RES116137 (Other: Case Western Reserve University)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: heart failure; congestive heart failure; telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health Guide using AHA protocols (Experimental): Participants in the study will receive the use of the Intel Health Guide, a telehealth device, with AHA customized heart failure protocols, response algorithms and educational content. Participants interact with the Intel Health Guide device, receiving immediate feedback when transmitting vitals measures and health question responses to a site monitored by their nurse case managers. Nurse case managers review and address concerns raised in vitals and/or question responses through standard care protocols established by their institution. Nurse case managers strive to enhance the participants quality of life, support continuity of care, facilitate provision of services in the appropriate setting to promote positive health outcomes.
  Interventions: Device: Health Guide using AHA heart failure protocols and content

INTERVENTIONS:
Device: Health Guide using AHA heart failure protocols and content — Participants in the study will receive the use of the Intel Health Guide, a telehealth device, with AHA customized heart failure protocols, response algorithms and educational content. Participants interact with the Intel Health Guide device, receiving immediate feedback when transmitting vitals measures and health question responses to a site monitored by their nurse case managers. Nurse case managers review and address concerns raised in vitals and/or question responses through standard care protocols established by their institution. Nurse case managers strive to enhance the participants quality of life, support continuity of care, facilitate provision of services in the appropriate setting to promote positive health outcomes.
  Other Names: Intel Health Guide

SUMMARY:
This purposed of this study is to ascertain if the implementation of remote patient management systems utilizing American Heart Association (AHA) guideline-based heart failure protocols and educational content can improve the management of patients with congestive heart failure.

DETAILED DESCRIPTION:
This prospective, comparative study uses a pre-post test design to ascertain if the implementation of remote patient management systems utilizing AHA guideline-based heart failure protocols and educational content can successfully address the following objectives:

* validate the suitability of the Intel Health Guide to deploy AHA guideline-based patient care protocols and health content to patients managing congestive heart failure
* confirm that the AHA protocols as deployed on the HGS are supportive for clinicians following the AHA guidelines in a telehealth environment
* validate and verify that the data intended to be collected was effectively collected
* measure patient and provider satisfaction with use of the system

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of Heart Failure NYHA and is currently in functional class II- IV status.
* Patient has been hospitalized for an episode of acute HF decompensation within the last 30 days.
* Patients with other co-morbidities such as atrial fibrillation, diabetes, coronary artery disease, COPD, hypertension, may be included in this evaluation. These conditions shall be documented during enrollment.
* Have telephone line or broadband internet availability to connect Intel® Health Guide.
* Are physically and mentally capable to complete the monitoring process or have a caregiver capable of assisting in the use of the Intel® Health Guide.
* Will be willing and able to sign an informed consent form to participate in this evaluation for a duration of 60 days.
* Live within a reasonable distance (30 miles or less) from the institution.

Exclusion Criteria:

* Have a life expectancy of less than six months.
* Live in a nursing home or other multi-member assisted living facility.
* Intend to be away from their home for more than 2 weeks (14 days) total during the 60 days.
* Are unable to read English at a minimum 5th grade level.
* Do not live within a reasonable distance (30 miles or less) from the institution.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George E Kikano, MD, CPE, Principal Investigator — Chair, Dept. of Family Medicine, Case Western Reserve University/University Hospitals; Ileana L Piña, MD, MPH, Principal Investigator — Professor, Medicine & Epi/Biostats, Case Western Reserve University/University Hospitals
Locations (1):
- University Hospitals Home Care Services, Warrensville Heights, Ohio, United States

REFERENCES:
- See also: The American Heart Association's mission is to build healthier lives, free of cardiovascular diseases and stroke. — http://www.heart.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The University Hospitals Home Care Services program, which is nurse driven for patients within a certain radius from the hospital, was the source of patient referral. Patients were self-selected and consented following hospital discharge with a heart failure diagnosis, were home bound, thus qualified for the home care nursing program.
Period: Overall Study
Arm/Group | Health Guide Using AHA Protocols
Started | 26
Completed | 25
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Health Guide Using AHA Protocols
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Participants Measured Vitals and Completed Protocol Sessions
Description: Measuring the percentage of available days the patient measures and records his/her vitals (weight, blood pressure, blood oxygen saturation level, glucose level) and completes his/her protocol sessions during the monitoring period. Utility was defined as days of activity and interaction of the patient with the monitor / days of actual monitoring possible.
Time Frame: 60 days
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Health Guide Using AHA Protocols
Number analyzed (Participants) | 26
percentage of days | 88 [82.2 to 96.9]

2. Primary Outcome: Percentage of Health Sessions That Patients Measured and Recorded Vitals
Description: Measuring the percentage of available health sessions that the patient measures and records his/her vitals (weight, blood pressure, blood oxygen saturation level, glucose level) and during the monitoring period. Adherence (or patient compliance) was defined as the percent of actual completed sessions from the number of scheduled sessions offered.
Time Frame: 60 days
Measure: Mean (Full Range); unit: percentage of health sessions completed
Arm/Group | Health Guide Using AHA Protocols
Number analyzed (Participants) | 26
percentage of health sessions completed | 77 [67.4 to 97.2]

3. Secondary Outcome: Patient Quality of Life Using the Kansas City Cardiomyopathy Questionnaire (KCCQ) Mean Clinical Summary Score Change
Description: Impact of the Intel® Health Guide System using AHA heart failure protocols and educational content on the patient's quality of life as measured pre and post intervention (mean clinical summary score change) using the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is a 23-item self-administered questionnaire used to measure the patient's perception of their health status. The KCCQ tool quantifies six (6) distinct domains (symptom, physical function, quality of life, social limitation, self-efficacy and symptom stability) and two (2) summary scores (clinical and overall). This measure represents the Mean Clinical Summary Score Change.
Time Frame: Baseline is taken at the beginning of the study, 2nd is at 30 days and 3rd is at 60 days.
Population: The scale is from 0 to 100; 100 being the best quality of life. A change of 5 points or higher is clinically significant. The first five items (physical limitation, symptom stability, symptom frequency, total symptom score) are combined with the quality of life domain to get the clinical score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Guide Using AHA Protocols
Number analyzed (Participants) | 26
score on a scale
  Baseline | 50.74 (22.89)
  Second | 51.69 (22.95)
  Third | 65.36 (22.06)

4. Secondary Outcome: Patient Quality of Life Using the Kansas City Cardiomyopathy Questionnaire (KCCQ) Mean Overall Score Change
Description: Impact of the Intel® Health Guide System using AHA heart failure protocols and educational content on the patient's quality of life measured pre and post intervention (mean overall score change) using the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is a 23-item self-administered questionnaire used to measure the patient's perception of their health status. The KCCQ tool quantifies six (6) distinct domains (symptom, physical function, quality of life, social limitation, self-efficacy and symptom stability) and two (2) summary scores (clinical and overall). This measure represents the Mean Overall Score Change.
Time Frame: Baseline is at the beginning of study, 2nd is at 30 days and 3rd is at 60 days.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Guide Using AHA Protocols
Number analyzed (Participants) | 26
score on a scale
  Baseline | 48.74 (25.06)
  Second | 49.84 (25.18)
  Third | 63.38 (26.28)

ADVERSE EVENTS:
Time Frame: 60 days from consent and enrollment
Arm/Group | Health Guide Using AHA Protocols
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 13/26
Other Adverse Events (participants affected / at risk) | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Guide Using AHA Protocols (N=26)
Rehospitalization (Cardiac disorders) | 4 (4) — Patients hospitalized due to heart failure complications
Rehospitalization (General disorders) | 9 (9) — Rehospitalization fore reasons other than heart failure.

LIMITATIONS AND CAVEATS:
Limitations of this study due to funding limitations included: very small patient sample size (26) from a single center enrollment in Northeast Ohio, with a short monitoring period (60 days), non-randomized and with no control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT01275846/Prot_SAP_000.pdf